CLINICAL TRIAL: NCT04274023
Title: Phase II Study on TSR-042 in Advanced Clear Cell Sarcoma
Brief Title: Study on TSR-042 in Advanced Clear Cell Sarcoma
Acronym: ACCeSs
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty of enrollment
Sponsor: Italian Sarcoma Group (Network)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISG-ACCeSs
Record Dates: First submitted 2020-02-13; First posted 2020-02-18 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Sarcoma, Clear Cell
Keywords: advanced clear cell sarcoma; anti-PDL1
MeSH Terms: conditions — Sarcoma, Clear Cell | interventions — dostarlimab

STUDY DESIGN:
Intervention Model Description: Single arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TSR-042 arm (Experimental): TSR-042 at a dose of 500 mg in IV infusion (given over t30-minutes) every 21 days for the first 4 doses, followed by 1.000 mg on day 1 of every 42 day.
  Interventions: Drug: TSR-042

INTERVENTIONS:
Drug: TSR-042 — TSR-042 is an IgG4 humanized monoclonal antibody that binds with high affinity to PD-1, resulting in inhibition of binding to PD-L1 and PD-L2.

SUMMARY:
Phase II,single arm study designed to explore the activity of TSR-042, an immunotherapy agent, in patients with a diagnosis of advanced or metastatic clear cell sarcoma (CCS).

DETAILED DESCRIPTION:
Phase II, single arm, not randomized, European multicentric study designed to explore the activity of TSR-042, a human monoclonal anti-PD-1 inhibitor, in a population of patients with a diagnosis of advanced/metastatic clear cell sarcoma (CCS).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Histological centrally confirmed diagnosis of clear cell sarcoma
3. Availability of archived tumor tissue block, or 15 slides.
4. Locally advanced disease
5. Measurable disease based on RECIST 1.1
6. Patient can be naive or previously treated with 1 or 2 systemic regimens given for recurrent and/or metastatic disease
7. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2
8. Adequate bone marrow function
9. Adequate organ function
10. Cardiac ejection fraction ≥50%
11. At least 18 years of age on day of signing informed consent.
12. Non-pregnant female patients
13. Non-ot breastfeed during the study for 90 days after the last dose of study treatment.
14. Male participant agrees to use an adequate method of contraception
15. No history of arterial and/or venous thromboembolic event within the previous 12 months.
16. Participant receiving corticosteroids may continue as long as their dose is stable for least 4 weeks prior to initiating protocol therapy.
17. Patients who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Participant must not be simultaneously enrolled in any interventional clinical trial
2. Previous treatment with any non-investigational agents within 14 days of first day of study drug dosing.
3. Must not have received investigational therapy ≤ 4 weeks, or within a time interval less than at least 5 half-lives of the investigational agent, whichever is shorter, prior initiating protocol therapy
4. Other primary malignancy with <5 years clinically assessed disease-free interval, except basal cell skin cancer, cervical carcinoma in situ, or other neoplasms judged to entail a low risk of relapse
5. Previous treatment with radiation therapy within 14 days of first day of study drug dosing, or patients who have not recovered from adverse events due to agents administered more than 4 weeks earlier
6. Has known active central nervous system (CNS) metastases, leptomeningeal metastases, and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable, have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability
7. Has active, non-infectious pneumonitis
8. Has an active infection requiring systemic therapy
9. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agents
10. Has received a live vaccine within 30 days of planned start of study therapy
11. Major surgery within 3 weeks prior to study entry
12. Any one of the following currently or in the previous 6 months:

Myocardial infarction, congenital long QT syndrome, Torsades de Pointes, arrhythmias right bundle branch block and left anterior hemiblock unstable angina coronary/peripheral artery bypass graft, symptomatic congestive heart failure New York Heart Association Class III or IV, cerebrovascular accident, or transient ischemic attack symptomatic pulmonary embolism. Ongoing cardiac dysrhythmias of Grade >=3, atrial fibrillation of any grade,or QTcF interval >470 msec 14. Severe and/or uncontrolled medical disease 15. Patient experienced ≥ Grade 3 immune-related AE with prior immunotherapy 16. Participant has a diagnosis of immunodeficiency or has receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to initiating protocol therapy 17. Any known active hepatitis B or hepatitis C 18. Any known history of human immunodeficiency virus 19. Subjects who have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment) 20. Expected non-compliance to medical regimens 21. Known history of interstitial lung disease 22. Active autoimmune disease that has required systemic treatment in the past 2 years 23. Known severe hypersensitivity reactions to monoclonal antibodies, any history of anaphylaxis, or uncontrolled asthma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-01-29 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | At week 12
  Response rate according Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

SECONDARY OUTCOMES:
Immune-related RECIST (ir-RECIST) response rate | At weeks 6, 12, 24, 36, 48, 60, 72, 84, 96
  Response rate according ir-RECIST criteria
Choi criteria response rate | At weeks 6, 12, 24, 36, 48, 60, 72, 84, 96
  Response rate according Choi criteria
Progression Free Survival (PFS) | At 3 and 5 years
  Survival without disease progression
Overall Survival | At 3 and 5 years
  Proportion of patients who are still alive at 36 and 60 months after have started the treatment
Clinical Benefit Rate | Month 6
  Proportion of patients who experienced Complete Response, Progression Response or Stable Disease for over 6 months
Adverse events related to the treatment | Week 3, week 6, week 9, week 12, week 18, week 24, week 36, week 48, week 60, week 72
  Safety in term of grading of adverse event is evaluate from the firs treatment dose throughout the study according to CTCAE 5.0
Growth Modulation Index (GMI) | At weeks 6, 12, 24, 36, 48, 60, 72, 84, 96
  Correlation between response and prior disease medical treatment: ratio of time to progression with the nth line of therapy to the those with the n-1th line.
Quality of Life according the 30 questions European Organization for Research and Treatment of Cancer Quality of Life Questionnaire | Day1 Cycle 2, Day 1 Cycle 3, Every 3 cycles (Day1Cyle6, Day1Cycle 9, …) and through study completion, an average of 1 year
  Evaluation of the quality of life collected with European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30
Quality of Life according the questionnaire Euro Quality Of Life 5 Domains (EQ-5D) | Day1 Cycle 2, Day 1 Cycle 3, Every 3 cycles (Day1Cyle6, Day1Cycle 9, …) and through study completion, an average of 1 year
  Evaluation of the quality of life collected with Euro Quality Of Life 5 Domains (EQ-5D)
Safety according the Patient Reported Outcome according Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Day1 Cycle 2, Day 1 Cycle 3, Every 3 cycles (Day1Cyle6, Day1Cycle 9, …) and through study completion, an average of 1 year
  Evaluation of the quality of safety reported by the patient with the PRO-CTCAE

OTHER OUTCOMES:
Expression level of PD1 and PDL1 at pre-treatment evaluated on cancer cells and in tumor infiltrating myeloid cells | Day1 (pre-treatment)
  Analysis of immune contexture in pretreatment tumor tissue.
Frequency in the expression of myeloid-derived suppressor cells in peripheral blood mononuclear cell | Day1, day15, day45 of treatment and through study completion, an average of 1 year
  Immunological monitoring of peripheral blood immune subsets, to evaluate the systemic immunological status of patients,
Frequency in the expression of anti-tumor immune cells in PBMC collected at baseline and during TSR-042. | Day1, day15, day45 of treatment and through study completion, an average of 1 year
  Immunological monitoring of peripheral blood immune subsets, to evaluate the systemic immunological status of patients,

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Stacchiotti, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori di Milano
Locations (1):
- Fondazione IRCSS Istituto Nazionale dei Tumori, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Granter SR, Weilbaecher KN, Quigley C, Fletcher CD, Fisher DE. Clear cell sarcoma shows immunoreactivity for microphthalmia transcription factor: further evidence for melanocytic differentiation. Mod Pathol. 2001 Jan;14(1):6-9. doi: 10.1038/modpathol.3880249. PMID 11211309
- [Background] Antonescu CR, Tschernyavsky SJ, Woodruff JM, Jungbluth AA, Brennan MF, Ladanyi M. Molecular diagnosis of clear cell sarcoma: detection of EWS-ATF1 and MITF-M transcripts and histopathological and ultrastructural analysis of 12 cases. J Mol Diagn. 2002 Feb;4(1):44-52. doi: 10.1016/S1525-1578(10)60679-4. PMID 11826187
- [Background] Stacchiotti S, Grosso F, Negri T, Palassini E, Morosi C, Pilotti S, Gronchi A, Casali PG. Tumor response to sunitinib malate observed in clear-cell sarcoma. Ann Oncol. 2010 May;21(5):1130-1. doi: 10.1093/annonc/mdp611. Epub 2010 Jan 21. No abstract available. PMID 20093352
- [Background] Tazzari M, Palassini E, Vergani B, Villa A, Rini F, Negri T, Colombo C, Crippa F, Morosi C, Casali PG, Pilotti S, Stacchiotti S, Rivoltini L, Castelli C. Melan-A/MART-1 immunity in a EWS-ATF1 translocated clear cell sarcoma patient treated with sunitinib: a case report. BMC Cancer. 2015 Feb 14;15:58. doi: 10.1186/s12885-015-1044-0. PMID 25880253